CLINICAL TRIAL: NCT02149927
Title: Neural Mechanisms of Sevoflurane Induced Anesthesia: an EEG fMRI Study in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 56012/12
Record Dates: First submitted 2014-04-22; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Anesthesia; Drug Effects
Keywords: EEG; fMRI; connectivity; sevoflurane
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sevoflurane (Experimental): Single arm: dose escalation of study medication
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane

SUMMARY:
In imaging functional connectivity (FC) analyses of the resting brain, alterations of FC during unconsciousness have been reported. These results are in accordance to recent electroencephalographic studies observing impaired top-down processing during anesthesia. In this study, simultaneous records of functional magnetic resonance imaging (fMRI) and electroencephalogram (EEG) were performed to investigate the causality of neural mechanisms during sevoflurane anesthesia by correlating FC in fMRI and directional connectivity (DC) in electroencephalogram.

ELIGIBILITY:
Inclusion Criteria:

* ASA I
* male
* age > 18y

Exclusion Criteria:

* drug abuse
* history of psychiatric or neurologic diseases
* amblyacousia, deafness
* contradictions to the study drug (sevoflurane)
* implants
* piercings, tatoos

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes of information processing (entropy) in EEG and functional connectivity (BOLD ICA and small group network architecture) in fMRI during sevoflurane anesthesia at states awake, 2vol%, 3vol% and EEG endpoint burst suppression | 10 minutes for each condition
  Changes of fMRI functional connectivity and of EEG information processing during different levels of sevoflurane anesthesia from wakefulness to deep anesthesia:
  At each anesthetic level at equilibrated states awake, 2vol%, 3vol% and EEG endpoint burst suppression, EEG and fMRI are recorded simultaneously for about 10 minutes. For each level EEG and fMRI connectivity analysis are performed using the recording length of 10 minutes. This results in one outcome parameter for EEG and fMRI connectivity. Furthermore, both modalities are combined resulting in one combined parameter for each level.
  For EEG analysis permutation entropy as a measure of information content in EEG, and symbolic transfer entropy as a measure of directed interaction in EEG are used. fMRI functional connectivity analysis is based on BOLD ICA and on network analysis of the BOLD time series.

SECONDARY OUTCOMES:
Assessment of the brain network structure during recovery in EEG and fMRI | 10 minutes for each condition
  Identical technical setup than main outcome

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard F Kochs, MD, Study Chair — Klinikum rechts der Isar, Technische Universität München, Munich, Germany
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany